CLINICAL TRIAL: NCT05040061
Title: SkillJoy Randomized Controlled Trial: Testing a Smartphone Intervention for Anxiety and Reinforcement
Brief Title: SkillJoy Clinical Trial
Acronym: SkillJoy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Skidmore College (Other)
Collaborators: Penn State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2108-974
Record Dates: First submitted 2021-08-24; First posted 2021-09-10 (Actual); Last update posted 2021-09-10 (Actual); Status verified 2021-09

CONDITIONS: Generalized Anxiety Disorder
Keywords: Worry; Savoring; Ecological Momentary Intervention; Generalized Anxiety Disorder; Positive Emotion
MeSH Terms: conditions — Generalized Anxiety Disorder

STUDY DESIGN:
Intervention Model Description: Participants screened to select-in GAD with a clinical interview are randomly assigned to either a savoring treatment intervention condition (SkillJoy) or an active treatment control condition emphasizing self-monitoring.
Who Masked: Participant
Masking Description: Participant were not made aware of the existence of the condition to which they were not assigned, nor the nature of that condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SkillJoy Intervention (Experimental): The savoring treatment consisted of an ecological momentary intervention (EMI) for learning and practicing savoring skills-SkillJoy. SkillJoy prompted participants to attend to positive aspects of the present moment, plan and engage in enjoyable activities, record and reflect on positive experiences, note events that turned out well, and look forward to positive events.
  Interventions: Behavioral: SkillJoy Intervention
- Active Self-Monitoring Control Intervention (Active Comparator): The active self-monitoring control EMI consisted of similar activities, but they all omitted savoring practices. These activities included attending to any current thoughts and feelings, planning everyday activities, remembering and recording daily events, and anticipating important events.
  Interventions: Behavioral: Active Self-Monitoring Control Intervention

INTERVENTIONS:
Behavioral: SkillJoy Intervention — The savoring treatment consisted of an ecological momentary intervention (EMI) for learning and practicing savoring skills-SkillJoy. SkillJoy prompted participants to attend to positive aspects of the present moment, plan and engage in enjoyable activities, record and reflect on positive experiences, note events that turned out well, and look forward to positive events.
  Arms: SkillJoy Intervention
Behavioral: Active Self-Monitoring Control Intervention — The active self-monitoring control EMI prompted participants to notice and write current thoughts and feelings, plan the day's major activities, remember and write about their daily events, and anticipate upcoming important events.
  Arms: Active Self-Monitoring Control Intervention

SUMMARY:
This study is a randomized controlled trial comparing a smartphone-delivered savoring intervention (SkillJoy) for Generalized Anxiety Disorder to an active treatment control.

DETAILED DESCRIPTION:
The current study seeks to determine if the positivity intervention SkillJoy, a smartphone-based, ecological momentary intervention (EMI), can reduce worry and generalized anxiety disorder (GAD) symptoms, increase positive emotion and wellbeing, improve reinforcement and probabilistic learning, increase savoring and reduce kill-joy thinking, and decrease avoidance of negative emotional shifts relative to an active treatment control in a GAD sample. Skills for generating positive emotion may reduce symptoms and increase well-being for those with GAD. To test this approach, participants with GAD were randomly assigned to either a savoring treatment or a self-monitoring control.The savoring treatment consisted of an ecological momentary intervention (EMI) for learning and practicing savoring skills-SkillJoy. SkillJoy prompted participants to attend to positive aspects of the present moment, plan and engage in enjoyable activities, record and reflect on positive experiences, note events that turned out well, and look forward to positive events. The active self-monitoring control EMI consisted of similar activities, but they all omitted savoring practices. These activities included attending to any current thoughts and feelings, planning everyday activities, remembering and recording daily events, and anticipating important events. Both EMIs were delivered by apps on participants' smartphones for seven days with 30th day follow-up. Secondarily, the current study will assess differences between those with GAD and non-anxious controls on a computerized probabilistic reinforcement learning task and baseline savoring questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Meet clinical criteria for Generalized Anxiety Disorder on the GAD-Q-IV and the GAD section of the Mini-International Neuropsychiatric Interview (MINI).
* Must be at least 18 years old to participate.
* Pregnant women will be allowed to participate.

Exclusion Criteria:

* They do not meet criteria for GAD on the GAD-Q-IV and the INI or do not fall one standard deviation below the subject pool mean on the GAD-Q-IV (i.e., they fall between these two scores).
* They are younger than 18 years of age.
* They do not speak English.
* They are adults unable to consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2018-05-17 (Actual); Primary Completion 2019-12-07 (Actual); Study Completion 2019-12-07 (Actual)

PRIMARY OUTCOMES:
Pre- to Post-Trial and Pre-Trial to Follow-Up Change in The Penn State Worry Questionnaire | 8 day post-trial; 30th day follow-up
  A 16-item self-report scale of the severity and frequency of worry. Min. score of 16 and maximum score of 80. Decreases in scores suggest a better outcome.
Pre- to Post-Trial and Pre-Trial to Follow-Up Change in The Positive and Negative Affect Schedule, Expanded Form: Joviality Scale | 8 day post-trial; 30th day follow-up
  An 8-item measure of positive emotions. Min. score of 8 and maximum score of 40. Increases in scores suggest a better outcome.
Pre- to Post-Trial and Pre-Trial to Follow-Up Change in The Savoring the Moment Subscale of the Savoring Beliefs Inventory | 8 day post-trial; 30th day follow-up
  The SBI is a 14-item survey that measures beliefs about one's ability to savor. The savoring the moment subscale measures savoring of present-moment emotional experience. Min. score of 1 and maximum score of 7. Increases in scores suggest a better outcome.

SECONDARY OUTCOMES:
Pre- to Post-Trial and Pre-Trial to Follow-Up Change in Responses to Positive Affect Scale: Dampening Subscale | 8 day post-trial; 30th day follow-up
  Measure kill-joy thinking (a.k.a. "dampening"). Participants rated eight dampening items on a 5-point scale. Min. score of 8 and maximum score of 32. Decreases in scores suggest a better outcome.
Pre- to Post-Trial and Pre-Trial to Follow-Up Change in The Prioritizing Positivity Scale | 8 day post-trial; 30th day follow-up
  Measures the degree to which participants prioritized seeking positive experiences on six items with which participants either agree or disagree on a nine-point scale. Min. score of 6 and maximum score of 54. Increases in scores suggest a better outcome.
Pre- to Post-Trial and Pre-Trial to Follow-Up Change in The Life Orientation Test - Revised | 8 day post-trial; 30th day follow-up
  Measures optimism. It has 10 items rated on a four-point scale. Min. score of 6 and maximum score of 30. Increases in scores suggest a better outcome.
Pre- to Post-Trial and Pre-Trial to Follow-Up Change in The Beck Depression Inventory II | 8 day post-trial; 30th day follow-up
  A 21-item self-report survey that measures the presence and severity of depressive symptoms. Minimum score of 0 and maximum score of 63. Decreases in scores suggest a better outcome.
Pre- to Post-Trial and Pre-Trial to Follow-Up Change in Contrast Avoidance Questionnaire - Worry | 5 day mid-trial; 8 day post-trial; 30th day follow-up
  Measures frequency, severity, and motivation to use worry to cope with negative shifts in emotion and benefit from positive shifts in emotion. Min. score of 30 and maximum score of 150. Decreases in scores suggest a better outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Skidmore College, Saratoga Springs, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Any relevant de-identified IPD will be shared to other researchers upon reasonable, direct request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will be available at the time of reasonable request.
Access Criteria: Data will be provided to 1) trained and credentialed researchers who 2) make a direct request to the authors with 3) a clearly-stated rationale and purpose for receiving the data that is considered relatively reasonable by the authors (e.g., to re-analyze a published statistical analysis).

REFERENCES:
- [Derived] LaFreniere LS, Newman MG. Savoring changes novel positive mindset targets of GAD treatment: Optimism, prioritizing positivity, kill-joy thinking, and worry mediation. Behav Res Ther. 2024 Jun;177:104541. doi: 10.1016/j.brat.2024.104541. Epub 2024 Apr 16. PMID 38640622
- [Derived] LaFreniere LS, Newman MG. Upregulating positive emotion in generalized anxiety disorder: A randomized controlled trial of the SkillJoy ecological momentary intervention. J Consult Clin Psychol. 2023 Jun;91(6):381-387. doi: 10.1037/ccp0000794. Epub 2023 Jan 30. PMID 36716146

DOCUMENTS (3):
  • Study Protocol (2018-04-30): https://cdn.clinicaltrials.gov/large-docs/61/NCT05040061/Prot_000.pdf
  • Statistical Analysis Plan (2019-05-05): https://cdn.clinicaltrials.gov/large-docs/61/NCT05040061/SAP_001.pdf
  • Informed Consent Form (2016-02-22): https://cdn.clinicaltrials.gov/large-docs/61/NCT05040061/ICF_002.pdf